CLINICAL TRIAL: NCT01793350
Title: A Combined Phase 1 + 2 Clinical Trial Evaluating the Safety and Efficacy of BC-DN-01 in the Treatment of Painful Diabetic Peripheral Neuropathy
Brief Title: Safety and Efficacy Study of BC-DN-01 in Painful Diabetic Peripheral Neuropathy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioChemics, Inc. (Industry)
Collaborators: Harrison Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BC-222
Record Dates: First submitted 2013-02-05; First posted 2013-02-15 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Diabetic Neuropathy, Painful
Keywords: Diabetes; Mellitus; Painful; Neuropathy; Peripheral
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BC-DN-01 topically applied cream, DPN (Active Comparator): 4g topically applied BC-DN-01 cream applied twice daily to each leg and foot, for 12 weeks
  Interventions: Drug: BC-DN-01 topically applied cream
- Placebo topically applied cream, DPN (Placebo Comparator): 4g topically applied cream applied twice daily to each leg and foot, for 12 weeks

INTERVENTIONS:
Drug: BC-DN-01 topically applied cream — Phase 1 - week 1 - total daily dose 160mg benfotiamine as 8g BC-DN-01 Phase 1 - week 2 - total daily dose 320mg benfotiamine as 16g BC-DN-01 Phase 2 - for 12 weeks - total daily dose 320mg benfotiamine as 16g BC-DN-01
  Other Names: active ingredient of BC-DN-01 : benfotiamine
  Arms: BC-DN-01 topically applied cream, DPN

SUMMARY:
A combined Phase 1 & 2 study to evaluate the safety and effectiveness of a new diabetic neuropathy topical cream, containing benfotiamine, will be performed at 5 clinical sites and plans for BC-DN-01 administration in up to 135 volunteer patients using a standard Phase 1 + 2 design. Up to 15 subjects will receive BC-DN-01 in Study Phase 1 and up to 120 subjects will receive BC-DN-01 or placebo in Study Phase 2.

In Phase 1, a BC-DN-01 dose delivering 160mg benfotiamine/day (80mg twice daily) will be administered for the first 7 days. On visit day 0, patients will commence study treatment. Patients will be interviewed by phone on day 3 and return to clinic on day 7 for safety assessments. If the drug is well-tolerated and no significant adverse events experienced, the total daily BC-DN-01 dose will be increased on days 7-14 to 320mg benfotiamine/day (160mg b.i.d.). Patients will be interviewed by telephone on day 10 and return to clinic on day 14 for safety assessments.

Once the safety profile has been determined in Phase 1 as acceptable, the Phase 2 study will be initiated to evaluate clinical efficacy of BC-DN-01. Phase 2 is a randomized, placebo-controlled, double-blind, parallel study. Participants receive placebo or BC-DN-01 based on 1:1 randomization. Each patient will apply 4g of the study medication to each leg twice-a-day administering 320mg benfotiamine dose/day for 12 weeks.

Participants will be evaluated in the clinic at baseline and at 4, 8, and 12-week time points; study staff will interview the patients by telephone on weeks 2, 6, and 10.

The primary endpoint of the phase 2 trial is reduction in DPN pain measured by the Brief Pain Inventory. Phase 2 patients will be invited to give written consent to take part in biopsy sampling and additional gene expression analysis.

DETAILED DESCRIPTION:
The study will be performed at 5 clinical sites and plans for BC-DN-01 administration in up to 135 volunteer patients using a standard Phase 1 + 2 design. Based on conservative but approximate drop-out estimates of 20% in Study Phase 1 and 30% in Study Phase 2, up to 15 subjects will receive BC-DN-01 in Study Phase 1 and up to 120 subjects will receive either BC-DN-01 or placebo in Study Phase 2. It is anticipated that the enrolment of 135 subjects will allow for 12 and 84 evaluable in Study Parts 1 and 2, respectively.

Patient screening for study eligibility, randomisation, treatment administration, and safety and efficacy evaluations will be conducted at clinic visits in a qualified clinical research facility. It is anticipated that up to fifteen patients will be enrolled in the Phase 1 portion of the study intended to evaluate the safety and tolerability of daily, escalating doses of BC-DN-01 for two weeks. This portion of the study is not blinded and non-randomized. Upon completion of Phase 1, results will be used for the decision to initiate the Phase 2 portion of the study. It is anticipated that up to one hundred twenty (120) patients will be enrolled in Phase 2 and randomized to receive either placebo or a fixed BC-DN-01 dose for twelve weeks. Phase 2 will be double-blind to minimize bias.

All clinical safety measurements, observations, reported adverse symptoms, and laboratory safety data for each patient will be reviewed and clinically relevant findings reported to the Data Safety Monitoring Board (DSMB) at the end of the Phase 1 and the end of the Phase 2 trials. The decision to continue trial conduct will be made by BioChemics, Inc., and may be based on recommendations provided by a study continuation/study termination opinion by the DSMB. At no time will individual patient data or commentary thereon, from the blinded Phase 2 portion of the trial be shared by the DSMB with BioChemics, Inc. personnel or their study conduct partners.

This study is not formally powered to test a statistical hypothesis. The primary objective is to determine the magnitude of pain relief following a daily administration of 16g BC-DN-01 (320mg benfotiamine) compared to Placebo (Phase 2). This value will be used to determine the sample size needed in future clinical trials to ensure adequate analytical power to demonstrate efficacy.

Phase 1

Patients considered eligible for enrolment to the phase 1 study will be required to comply will all of the inclusion and exclusion criteria, including:

* Consented to phase 1 trial participation
* Met the protocol criteria for inclusion and exclusion (except inc criterion #8, #9 and exc criteria #3))
* Have not taken neuropathy pain medication for at least 2 weeks

Visit 1 (Screening) After providing written informed consent patients will undergo a physical examination, including leg and feet assessment, vital signs measured and safety blood samples taken including serum pregnancy test for women of child bearing potential.

Visit 2 (Baseline - Day 0) Patients will undergo a physical examination, including leg and feet assessment, vital signs measured and safety blood samples taken including urine pregnancy test for women of child bearing potential.

Patients will be dispensed BC-DN-01 study medication to provide 1 week of treatment, of 2g doses per leg, twice daily giving a total dose of 160mg benfotiamine/day (80mg b.i.d.). The first dose will be given by the study nurse, to demonstrate the correct way to apply the cream.

If the drug is well-tolerated and no significant adverse events are experienced, the total daily body BC-DN-01 dose will be increased following the clinic visit on day 7 (with the first increased dose of 160mg being applied on the evening of day 7)and then twice daily up to day 14, to 320mg benfotiamine/day (160mg b.i.d.).

Visit 3 (Day 7) Patients will undergo a leg and feet assessment, vital signs measured and safety blood samples taken including urine pregnancy test for women of child bearing potential.

Patients will be dispensed BC-DN-01 study medication to provide 1 week of treatment, of 4g doses per leg, twice daily.

Visit 4 (Day 14) Patients will undergo a physical examination, including leg and feet assessment, vital signs measured and safety blood samples taken including urine pregnancy test for women of child bearing potential. Patients will be contacted on days 3, 10 and 21-28 by telephone to be interviewed to discuss the medication, general health and any adverse events since the last clinic visit.

Phase 2

Once the safety profile has been determined in Phase 1 and considered acceptable, the Phase 2 study will be initiated to evaluate clinical efficacy of BC-DN-01. Patients participating in the Phase 1 safety evaluation may also participate in the randomised Phase 2 portion of the trial, at least four (4) months after completing the phase 1 trial. At that time, those patients, will be required to comply will all of the inclusion and exclusion criteria, including:

* Consented to phase 2 trial participation
* Met the protocol criteria for inclusion and exclusion
* Have not taken neuropathy pain medication for at least 2 weeks

Phase 2 is a randomised, placebo-controlled, double-blind, parallel study in up to 120 patients. Study participants will receive either placebo or BC-DN-01 based on 1:1 randomisation (at least 42 evaluable patients per treatment arm). Each volunteer patient will apply 4g of the study medication to each leg twice-a-day administering 320mg benfotiamine dose/day for 12 weeks.

The primary endpoint of the phase 2 trial is the reduction in pain level associated with DPN as measured by the Brief Pain Inventory (BPI). The duration of pain reduction will also be assessed.

The secondary efficacy endpoints include the evaluation of Sural and Peroneal motor nerve conduction velocities, Neuropathy Symptom Score, Neuropathy Disability Score, , Intra-epidermal nerve fibre density in the legs of these patients, hyperaesthesia and changes in lack of sensation in the leg and foot. Xerosis and changes in diabetes-related skin pathology, such as infiltration by inflammatory cells and mast cell degranulation as well as changes in the gene expression profiles of these tissues will also be assessed.

Visit 1 (Screening) After providing written informed consent patients will undergo a physical examination, including leg and feet assessment, vital signs measured and safety blood samples taken including serum pregnancy test for women of child bearing potential.

Visit 2 (Baseline - Day 0) Patients will undergo a physical examination, including leg and feet assessment, vital signs measured and safety blood samples taken including urine pregnancy test for women of child bearing potential.

Patients will be randomised to a 50:50 BC-DN-01:placebo arm and dispensed study medication to provide 4 weeks of treatment, of 4g doses per leg, twice daily giving the equivalent total dose of 320mg benfotiamine/day (80mg b.i.d.). The first dose of study medication will be given by the study nurse, to demonstrate the correct way to apply the cream.

Visits 3 (Week 4) 4 (Week 8) and 5 (Week 12) Patients will undergo a leg and feet assessment, vital signs measured and safety blood samples taken including urine pregnancy test for women of child bearing potential.

Patients will be asked to complete questionnaires regarding DPN pain, sensory tests and visual assessments of the skin on your legs and feet will be made Patients will undergo a nerve conduction velocity test, which tests how fast electrical signals move through the nerves on the leg.

Patients will be contacted on weeks 2, 6, 10 and 14 by telephone to be interviewed to discuss the medication, general health and any adverse events since the last clinic visit.

ELIGIBILITY:
Inclusion Criteria:

1. Current diagnosis of Type I or II diabetes mellitus according to the American Diabetes Association Criteria of FPG≥ 7.0 mmol/l (126 mg/dl)
2. A current or historical reading of HbA1c 6.5-11%, using a test performed in a clinical laboratory using a method that is NGSP certified and standardised to the DCCT assay.
3. Ability to understand the nature of the trial and willingness to participate, documented by written informed consent.
4. Willingness and ability to comply with the study protocol requirements for the duration of the study.
5. Males and females of any ethnic origin and ≥18 years of age.
6. Negative serum pregnancy test at screening and a negative urine pregnancy test at randomisation, for women of childbearing potential only and assurance from the patient (males and females) of using satisfactory contraception methods (refer to section 4.9.6).
7. If on anti-diabetic medication, must have been on a stable therapeutic regimen for at least 30 days prior to randomisation.
8. Phase 2 - Peroneal Motor Nerve Conduction Velocity measurements 30-40 m/s. indicating a mild to moderate case of diabetic peripheral neuropathy
9. Phase 2 - Scores on the Brief Pain Inventory of ≥4.
10. An ability to apply topical medication to both legs from the knee to the toes, either by themselves or have a documentation of an assistant or partner to help with the administration of the trial drug product twice a day for the 12-week treatment period.
11. Patient must be willing to sign a Consent form to participate in this clinical trial.
12. Patient must be willing to sign a consent form to be sent to their primary physician to inform that the patient will stop taking disallowed concomitant medications prescribed by the physician.

    -

Exclusion Criteria:

1. Participation in any investigational drug study within 4 months preceding randomisation of this study.
2. Pregnancy, lactation, fertility without adequate protection against pregnancy (refer to section 4.9.6).

   1. A serum pregnancy test will be performed for women of childbearing potential with the haematological and clinical chemistry evaluations at screening and a urine pregnancy test immediately prior to randomisation.
   2. If the patient becomes pregnant during the study, the patient's participation in the remainder of the study will be terminated.
3. Phase 2 - Severe neuropathy (PMNCV < 30 m/s, prior amputations at the foot level and Charcot disease).
4. Current severe peripheral arterial disease requiring surgical intervention (however patients with previous successful intervention 12 weeks or more prior to randomisation will be eligible for the study (See Section 4.2.2.1 Peripheral Arterial Disease Determination).
5. End stage renal failure requiring dialysis or renal transplantation and patients who are expected to receive dialysis or transplantation in the near future should be excluded from the study.
6. Presence of any serious disease, including those of hepatic, hematologic, neurologic, or immune origin or an active malignant disease, which in the opinion of the investigator would affect response to pain relief treatment.
7. Presence of peripheral pain not associated with DPN, mono-neuropathies or proximal neuropathies, or central pain, which in the opinion of the investigator would affect response to pain relief treatment.
8. Presence of a medical condition diagnosed with other known causes of non-Diabetic Peripheral Neuropathy.
9. Known to be currently abusing alcohol or drugs.
10. Presence of acute skin disease or infection such as erysipelas and vasculitis of the lower extremities.
11. Current oral or topical use of benfotiamine or BC-DN-01 products.
12. Hypersensitivity to benfotiamine or any component of BC-DN-01.
13. Concurrent administration or use of Lyrica, Cymbalta, or capsaicin use within the 2 weeks prior to randomisation (see Appendix 12.3 for full list of disallowed concomitant medications).
14. Any factors which, in the opinion of the investigator, will affect the patient's ability to safely participate in the study and meet study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of BC-DN-01 | 120 days
  The primary objective of this study is to assess the magnitude and duration of pain relief resulting from a fixed dose of BC-DN-01, compared to placebo, in patients with painful DPN as measured by the Brief Pain Inventory (BPI).

SECONDARY OUTCOMES:
Safety of BC-DN-01 | 120 days
  The secondary objectives for this study include assessing the safety and tolerability of 160mg b.i.d. of benfotiamine and determining the number of participants with adverse events as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Solomon Tesfaye, MD, FRCP, Principal Investigator — Royal Hallamshire Hospital, Sheffield, England
Locations (5):
- United Kingdom (5):
  - Royal Hallamshire Hospital, Sheffield, South Yorkshire
  - Ipswich Hospital, Ipswich, Suffolk
  - Birmingham Heartlands Hospital, Birmingham, West Midlands
  - MAC Clinical Research, Manchester
  - Manchester Royal Infirmary, Manchester